CLINICAL TRIAL: NCT02897141
Title: Use of mHealth Technology for Supporting Symptom Management in Underserved Persons Living With HIV
Brief Title: mVIP (Use of mHealth Technology for Supporting Symptom Management in Underserved Persons Living With HIV)
Acronym: mVIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Assistant Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAP1258; R21HS023963 (AHRQ)
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV; Health Management App; HIV symptoms
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mVIP group (Experimental): This group will receive targeted symptom strategies via a Health Management App developed from the UCSF symptom management manual based on the symptoms that they report. This is the intervention app group.
  Interventions: Device: Health Management App with symptom strategies
- Attention Control Group (Placebo Comparator): This group will received an app without symptom strategies, pre-loaded on their smartphones. This is the control app group.
  Interventions: Device: Control App

INTERVENTIONS:
Device: Health Management App with symptom strategies — The mVIP group will receive a Health Management App with symptom strategies. A mobile app which includes symptom strategies from the UCSF symptom management manual.
  Arms: mVIP group
Device: Control App — The attention control group will receive an app which asked them about their symptoms but did not provide symptoms strategies
  Arms: Attention Control Group

SUMMARY:
The goal of this study is to facilitate the dissemination and implementation of patient centered outcomes research using mHealth technology to improve self-management of adverse symptoms in persons living with HIV/AIDS (PLWH). Symptom management in PLWH is especially important because the US HIV epidemic continues to exact a huge toll, especially among Agency for Healthcare Research and Quality (AHRQ) priority populations including racial, ethnic, and sexual minorities and low-income persons. The incorporation of HIV symptom management strategies into patients' lives through the use of mHealth technologies has the potential to advance the effective dissemination and implementation of patient centered outcomes research findings.

DETAILED DESCRIPTION:
HIV has changed from an acute illness to a chronic disease. The success of HIV medications and treatments has significantly altered the course of the disease. While AIDS-related illnesses are no longer the primary threat, a new set of HIV-associated complications have emerged, resulting in a chronic disease that for many will span several decades of life. The ability to self-manage adverse symptoms of HIV illness has been shown to improve patient-centered outcomes. In response to this need, a team at University of California, San Francisco (UCSF) developed a paper-based symptom management manual with self-management strategies for 21 common HIV/AIDS adverse symptoms (PCOR evidence). The efficacy of the manual was demonstrated in a 775-person randomized controlled trial (RCT) over three months at 12 sites. However, subsequent use of these strategies has been very limited; mHealth offers an ideal platform for the implementation and dissemination of evidence-based strategies for HIV symptom management. Due to the high incidence of HIV among racial and ethnic minority populations, it is appropriate to develop mHealth tools tailored to the needs of these populations. mHealth technology has the potential to address many of the healthcare needs of persons living with HIV/AIDS (PLWH) including symptom management. In response to these current issues, this study seeks to inform the development and testing of a mHealth application that will incorporate findings from PCOR studies to improve the outcomes of PLWH. To improve outcomes for those most in need, study activities are focused on communities with the greatest burden of HIV in the US, including racial and ethnic minorities and those of low socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with HIV/AIDS
2. Over the age of 18 years
3. Able to provide written informed consent
4. Able to communicate in English
5. Health literacy level of marginal or inadequate (as measured by the Newest Vital Sign (NVS): total score of 3 or lower)
6. Report at least 2 HIV related adverse symptoms in the past week
7. Owner of a smart phone/tablet.

Exclusion Criteria:

1. Inability to communicate in English
2. Documented diagnosis of dementia
3. Pregnancy
4. Unable to understand consent procedure
5. Self-reporting no adverse symptoms within the past week. (HIV-related symptoms include: anxiety, constipation, cough, depression, diarrhea, dizziness, fever, forgetfulness, fatigue, nausea, night sweats, neuropathy, shortness of breath, dermatitis, swelling of arms, hand, legs, feet, insomnia, weight loss, oral thrush, and vaginal itching, burning and discharge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, RN-BC, FAAN, Principal Investigator — Columbia University
Locations (1):
- Columbia University School for Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- mVIP Group: This group will receive targeted symptom strategies from the University of California, San Francisco (UCSF) symptom management manual based on the symptoms that they report.
  Health Management App with symptom strategies: The mVIP group will receive a Health Management App with symptom strategies. A mobile app which includes symptom strategies from the UCSF symptom management manual.
- Attention Control Group: This group will have the Health Management App without symptom strategies pre-loaded on their smartphones.
  Health Management App without symptom strategies: The attention control group will receive the Health Management App preloaded on their smartphones without symptoms strategies
Period: Overall Study
Arm/Group | mVIP Group | Attention Control Group
Started | 40 | 40
Completed | 38 | 39
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- mVIP Group: This group will receive targeted symptom strategies from the UCSF symptom management manual based on the symptoms that they report.
  Health Management App with symptom strategies: The mVIP group will receive a Health Management App with symptom strategies. A mobile app which includes symptom strategies from the UCSF symptom management manual.
- Total: Total of all reporting groups
Arm/Group | mVIP Group | Attention Control Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.7) | 50.8 (9) | 50.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 15 | 23 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White, non-hispanic | 4 | 4 | 8
  Race: Black, non-hispanic | 29 | 26 | 55
  Race: Hispanic | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Education [Count of Participants; unit: Participants]
  Less than high school | 9 | 5 | 14
  High school | 11 | 14 | 25
  Some college or associates degree | 15 | 13 | 28
  Bachelors or advanced degree | 5 | 8 | 13
Annual income [Count of Participants; unit: Participants]
  Less than $10,000/year | 22 | 17 | 39
  $10,000-$19,999/year | 9 | 10 | 19
  $20,000-$59,999/year | 3 | 8 | 11
  Don't know or prefer not to answer | 6 | 5 | 11
Employment [Count of Participants; unit: Participants]
  Working (full, part, off-books) | 7 | 8 | 15
  Unemployed (looking, not looking) | 15 | 11 | 26
  Retired | 3 | 1 | 4
  Student | 2 | 2 | 4
  Disabled | 11 | 16 | 27
  Unspecified | 2 | 2 | 4
Antiretroviral therapy (ART) Use [Count of Participants; unit: Participants]
  None | 3 | 1 | 4
  2+ pills per day | 15 | 19 | 34
  1 pill per day | 21 | 20 | 41
  Prefer not to answer | 1 | 0 | 1
Virologically suppressed [Count of Participants; unit: Participants] | 34 | 34 | 68
Ever diagnosed with AIDS [Count of Participants; unit: Participants] | 17 | 24 | 41
Cluster of Differentiation 4 (CD4) count greater than 500 [Count of Participants; unit: Participants] | 22 | 20 | 42
Possible alcohol use disorder [Count of Participants; unit: Participants] | 15 | 10 | 25
Substance use weekly or more often [Count of Participants; unit: Participants] | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Status From Baseline to Week 12
Description: Change in Symptom Status calculates the difference in symptom scores between the intervention and control groups at baseline versus follow-up after 12 weeks. Symptom scores were determined using the Revised Sign and Symptom Check-List for HIV (SSC-HIVrev), where participants who reported experiencing any one of the 13 symptoms in the past 7 days were asked how much it bothered them (a little bit, somewhat, quite a bit, or very much). Instances where the symptom did not bother the individual were coded as "0" whereas instances where the symptom bothered the individual any amount were recoded as "1". The overall difference between groups at baseline and after 12 weeks ("difference of differences") falls within a range of -1 to 1, where lower numbers indicate the symptom bothered the person less, while higher numbers indicate it bothered them more. With the Difference Between Groups, a more negative score (closer to -1) represents a better outcome.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Intervention: Participants in the intervention group received self-care strategies for symptoms which they reported experiencing in the past seven days. Three self-care strategies were delivered for each reported symptom, along with short (3-27sec) videos to illustrate the strategy. At the end of the app session, participants were able to view a summary of their strategies.
- Control: Participants in the control group were asked the same questions about symptoms experienced in the last seven days (as dictated by the Revised Sign and Symptom Check-List for HIV -- SSC-HIVrev), though they were not given any self-care or symptom management strategies.
- Difference Between Groups: This represents the calculated difference between the average score changes from baseline to follow-up (12 weeks) among control and intervention group participants (described in the first two columns).
Arm/Group | Intervention | Control | Difference Between Groups
Number analyzed (Participants) | 40 | 40 | 80
score on a scale
  Anxiety | -0.858 (0.102) | -0.318 (0.118) | -0.541 (0.156)
  Cough of Shortness of Breath | -0.570 (0.105) | -0.421 (0.122) | -0.149 (0.161)
  Depression | -0.540 (0.106) | -0.007 (0.123) | -0.533 (0.163)
  Diarrhea | -0.240 (0.092) | -0.233 (0.107) | -0.007 (0.141)
  Difficulty falling asleep | -0.506 (0.106) | -0.433 (0.122) | -0.073 (0.162)
  Difficulty remembering | -0.343 (0.095) | -0.169 (0.110) | -0.174 (0.145)
  Dizziness | -0.319 (0.083) | -0.181 (0.095) | -0.138 (0.126)
  Fatigue | -0.566 (0.115) | -0.563 (0.132) | -0.003 (0.175)
  Fever, chills, sweats | -0.360 (0.086) | -0.084 (0.099) | -0.275 (0.132)
  Nausea or vomiting | -0.122 (0.066) | -0.185 (0.077) | 0.063 (0.101)
  Neuropathy | -0.713 (0.103) | -0.228 (0.119) | -0.485 (0.157)
  Skin problems | -0.219 (0.091) | -0.089 (0.105) | -0.130 (0.139)
  Weight loss or wasting | -0.254 (0.070) | -0.004 (0.081) | -0.250 (0.107)
Statistical Analysis 1: Comparison: Difference Between Groups; Anxiety; Test type: Superiority; p = 0.001, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.541, Standard Error of Mean 0.156
Statistical Analysis 2: Comparison: Difference Between Groups; Cough or Shortness of Breath; Test type: Superiority; p = 0.356, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count; a=0.05; Mean Difference (Final Values) = -0.149, Standard Error of Mean 0.161
Statistical Analysis 3: Comparison: Difference Between Groups; Depression; Test type: Superiority; p = 0.001, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.533, Standard Error of Mean 0.163
Statistical Analysis 4: Comparison: Difference Between Groups; Diarrhea; Test type: Superiority; p = 0.962, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -.007, Standard Error of Mean 0.141
Statistical Analysis 5: Comparison: Difference Between Groups; Difficulty falling or staying asleep; Test type: Superiority; p = 0.651, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.073, Standard Error of Mean 0.162
Statistical Analysis 6: Comparison: Difference Between Groups; Difficulty remembering; Test type: Superiority — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; p = 0.230, Mixed Models Analysis; Mean Difference (Final Values) = -0.174, Standard Error of Mean 0.145
Statistical Analysis 7: Comparison: Difference Between Groups; Dizziness; Test type: Superiority; p = 0.275, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.138, Standard Error of Mean 0.126
Statistical Analysis 8: Comparison: Difference Between Groups; Fatigue; Test type: Superiority; p = 0.987, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.003, Standard Error of Mean 0.175
Statistical Analysis 9: Comparison: Difference Between Groups; Fever, chills, sweats; Test type: Superiority; p = 0.037, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Net) = -0.275, Standard Error of Mean 0.132
Statistical Analysis 10: Comparison: Difference Between Groups; Nausea or vomiting; Test type: Superiority; p = 0.534, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 0.063, Standard Error of Mean 0.101
Statistical Analysis 11: Comparison: Difference Between Groups; Neuropathy; Test type: Superiority; p = 0.002, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.485, Standard Error of Mean 0.157
Statistical Analysis 12: Comparison: Difference Between Groups; Skin problems; Test type: Superiority; p = 0.349, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.130, Standard Error of Mean 0.139
Statistical Analysis 13: Comparison: Difference Between Groups; Weight loss or wasting; Test type: Superiority; p = 0.020, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.250, Standard Error of Mean 0.107

2. Secondary Outcome: Change in Quality of Life -- RAND-36
Description: 36-Item Short Form Survey (RAND-36) is a widely-used 36-item tool to measure health-related quality of life, where each item in the scale is scored as 0, 25, 50, 75, or 100. Scoring is a two-step process. First, precoded numeric values are recoded per the scoring key so that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores, where a lower score may indicate a better outcome for some of the scales, while it may indicate a better outcome for others.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: mVIP App participants
- Control: Control App participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 38 | 39
score on a scale
  Physical Functioning Scale | 66.22 (31.39) | 65.11 (28.97)
  Role limitations due to physical health scale | 55.41 (41.72) | 61.54 (41.30)
  Role limitations due to emotional problems scale | 62.16 (43.86) | 66.66 (41.43)
  Energy/fatigue scale | 51.35 (18.24) | 56.54 (19.67)
  Emotional well-being scale | 68.11 (15.42) | 73.23 (19.03)
  Social functioning scale | 66.89 (20.88) | 65.06 (26.47)
  Pain scale | 69.12 (20.41) | 63.14 (27.98)
  General health scale | 60.95 (21.34) | 60 (21.28)
  Physical health summary scale | 63.18 (23.80) | 63.03 (21.78)
  Mental health summary scale | 61.94 (18.53) | 65.83 (20.70)
Statistical Analysis 1: Comparison: Intervention vs Control; Physical functioning scale; Test type: Superiority — [Not specified]; p = 0.001, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; [Not specified]; Mean Difference (Final Values) = -3.06, Standard Error of Mean 7.27 — [Not specified]
Statistical Analysis 2: Comparison: Intervention vs Control; Role limitations due to physical health scale; Test type: Superiority — [Not specified]; p = 0.458, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; [Not specified]; Median Difference (Final Values) = 7.47, Standard Error of Mean 10.02 — [Not specified]
Statistical Analysis 3: Comparison: Intervention vs Control; Role limitations due to emotional problems scale; Test type: Superiority — [Not specified]; p = 0.725, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; [Not specified]; Mean Difference (Final Values) = 3.50, Standard Error of Mean 9.91 — [Not specified]
Statistical Analysis 4: Comparison: Intervention vs Control; Energy/fatigue scale; Test type: Superiority — [Not specified]; p = 0.807, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; [Not specified]; Mean Difference (Final Values) = -1.00, Standard Error of Mean 4.09 — [Not specified]; [Not specified]
Statistical Analysis 5: Comparison: Intervention vs Control; Emotional well-being scale; Test type: Superiority; p = 0.693, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 1.48, Standard Error of Mean 3.73
Statistical Analysis 6: Comparison: Intervention vs Control; Social functioning scale; Test type: Superiority; p = 0.128, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -8.93, Standard Error of Mean 5.80
Statistical Analysis 7: Comparison: Intervention vs Control; Pain scale; Test type: Superiority; p = 0.007, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -14.33, Standard Error of Mean 5.18
Statistical Analysis 8: Comparison: Intervention vs Control; General health scale; Test type: Superiority; p = 0.960, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.20, Standard Error of Mean 3.93
Statistical Analysis 9: Comparison: Intervention vs Control; Physical health summary scale; Test type: Superiority; p = 0.836, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.93, Standard Error of Mean 4.47
Statistical Analysis 10: Comparison: Intervention vs Control; Mental health summary scale; Test type: Superiority; p = 0.822, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.81, Standard Error of Mean 3.60

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29
Description: The PROMIS-29 includes seven health related quality of life domains on a 5-point scale from a score of 1 to 5 and the pain domain has two subdomains (interference and intensity) where pain intensity is assessed using a single 11-point numeric rating scale anchored between no pain (0) and worse imaginable pain (10). Raw scores are transformed using the T-score metric based on the item response theory calibrations in which scores have a mean of 50 and standard deviation of 10 for the general population in the US. T-scores can be estimated using the scoring tables listed in the PROMIS manuals. A higher PROMIS T-score implies more of the concept being measured; for instance, a higher PROMIS score on physical function indicates better functioning, whereas a higher score on depression indicates a greater severity of depression.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Intervention Arm: Participants received the mVIP App
- Control Arm: Participants received the control app
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 38 | 39
T-score
  Physical Function | 44.69 (9.09) | 45.70 (9.18)
  Anxiety | 55.85 (9.19) | 55.12 (10.56)
  Depression | 54.12 (10.46) | 50.53 (9.63)
  Fatigue | 51.76 (9.08) | 50.16 (9.89)
  Sleep Disturbance | 51.21 (9.64) | 52.85 (9.26)
  Satisfaction with participation in social roles | 48.86 (9.01) | 49.18 (8.72)
  Pain interference | 53.60 (7.90) | 53.25 (9.84)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Physical Function; Test type: Superiority; p = 0.529, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 0.79, Standard Error of Mean 1.25
Statistical Analysis 2: Comparison: Intervention Arm vs Control Arm; Anxiety; Test type: Superiority; p = 0.312, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 1.71, Standard Error of Mean 1.68
Statistical Analysis 3: Comparison: Intervention Arm vs Control Arm; Depression; Test type: Superiority; p = 0.841, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.36, Standard Error of Mean 1.81
Statistical Analysis 4: Comparison: Intervention Arm vs Control Arm; Fatigue; Test type: Superiority; p = 0.848, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 0.40, Standard Error of Mean 2.07
Statistical Analysis 5: Comparison: Intervention Arm vs Control Arm; Sleep Disturbance; Test type: Superiority; p = 0.208, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 2.58, Standard Error of Mean 2.03
Statistical Analysis 6: Comparison: Intervention Arm vs Control Arm; Satisfaction with participation in social roles; Test type: Superiority; p = 0.754, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 0.72, Standard Error of Mean 2.29
Statistical Analysis 7: Comparison: Intervention Arm vs Control Arm; Pain interference; Test type: Superiority; p = 0.454, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 1.25, Standard Error of Mean 1.66

4. Secondary Outcome: Engagement With Healthcare Provider
Description: Engagement with Health Care Provide scale is a 13-item scale in which subjects rate their interactions with their health care providers on a four-point scale with 1=always true and 4=never true in which a lower score indicates a better outcome. The scores are then collated to an aggregate score where the minimum value = 13 and the maximum value = 52. A low score indicates greater provider engagement, where as higher scores indicate lower provider engagement (less favorable outcome). The difference in scores at baseline and follow-up at three months was calculated within both the intervention and control groups, and the difference was then taken between the resulting means of those scores.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Arm: Participants received a control app
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 38 | 39
score on a scale | 16.65 (6.09) | 17.59 (7.56)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.252, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -2.52, Standard Error of Mean 2.19

5. Secondary Outcome: Medication Adherence
Description: Medication adherence was calculated by two scales: the Center for Adherence Support Evaluation (CASE) Adherence Index and the Visual Analogue Scale (VAS). The CASE Adherence Index consists of the composite scores of three questions evaluating self-reported measures of adherence. The minimum score on this scale is 3 while the maximum score on this scale is 16, with higher scores indicating better outcome. Scores greater than 10 indicate "good adherence," while scores less than or equal to 10 indicate poor adherence.
  The VAS asks subjects to indicate a point on a line that shows their best guess about how much of each drug they have taken from a scale of 0% to 100% in which 0% means they have taken no drug, 50% means they have taken half their drugs, and 100% means they have taken every single dose. Consequently, a higher score (100%) indicates
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Participants who received the mVIP app
- Control Arm: Participants who received the Control App
Arm/Group | Intervention | Control Arm
Number analyzed (Participants) | 38 | 39
score on a scale
  CASE adherence index | 12.97 (3.51) | 12.69 (3.00)
  Visual analogue scale | 85.97 (26.86) | 87.03 (20.56)
Statistical Analysis 1: Comparison: Intervention vs Control Arm; CASE adherence index; Test type: Superiority; p = 0.017, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -1.51, Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Intervention vs Control Arm; Visual analogue scale; Test type: Superiority; p = 0.338, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -4.88, Standard Error of Mean 5.06

6. Secondary Outcome: Health-IT Usability Evaluation Scale (Health-ITUES)
Description: Health Information Technology Usability Evaluation Scale (Health-ITUES) was used to measure usability. Health-ITUES consists of 20 items rated on a 5-point Likert scale from strongly disagree (score of 1) to strongly agree (score of 5) measuring actual usage, intention to use, satisfaction, perceived usefulness, perceived ease of use, perceived performance speed, learnability, competency, flexibility/customizability, memorability, error prevention, information needs, and other outcomes. A higher score (5) indicates higher usability. Overall score was calculated as the mean score from the score for quality of life, perceived usefulness, perceived ease of use, and user control.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Arm: Participants who received the mVIP app
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 38 | 39
score on a scale
  Overall | 4.39 (0.72) | 4.35 (0.63)
  Quality of Life | 4.50 (0.59) | 4.35 (0.78)
  Perceived usefulness | 4.23 (0.91) | 4.26 (0.74)
  Perceived ease of use | 4.64 (0.83) | 4.67 (0.71)
  User control | 4.32 (0.82) | 4.05 (0.93)
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Overall; Test type: Superiority; p = 0.743, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.07, Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Intervention Arm vs Control Arm; Quality of life; Test type: Superiority; p = 0.166, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.28, Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Intervention Arm vs Control Arm; Perceived usefulness; Test type: Superiority; p = 0.899, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = 0.03, Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Intervention Arm vs Control Arm; Perceived ease of use; Test type: Superiority; p = 0.803, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.07, Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Intervention Arm vs Control Arm; User Control; Test type: Superiority; p = 0.480, Mixed Models Analysis — Model controlled for age, sex, race, education, and CD4 count ; a=0.05; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.28

ADVERSE EVENTS:
Time Frame: Study duration, 12 weeks
Arm/Group | mVIP Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
Participants wanted reminders and login information sent via text instead of email. Both groups wanted summary reports of symptoms. Self-care strategy videos did not have sound. Generalizability is limited due to smartphone/tablet requirement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02897141/Prot_SAP_000.pdf